CLINICAL TRIAL: NCT02437435
Title: Effectiveness of Physiotherapy Treatment to Improve the Flow on Vascular Area of the Endometrial / Subendometrial in Uterus of Infertile Women With Hypoestrogenemia Evaluated by Three-dimensional Ultrasound Angiography.
Brief Title: Physiotherapy Treatment for Uterine Blood Flow Improved Dimensional Ultrasound Evaluated With Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Principal Investigator, César Gimilio, Physical Therapy, University of Valencia
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1406-VLC-044-CG-; 1406-VLC-044-CG (Other: Juana Crespo's Clinic)
Record Dates: First submitted 2015-04-15; First posted 2015-05-07 (Estimated); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Infertility
Keywords: assisted reproduction; physical therapy; manual therapy; uterine artery; Vascularization Index (VI); Doppler ultrasonography; vocal
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reproductive Technique Gimilio (Experimental): Patient supine, legs in triple flexion, feet on table, controlling legs left hand and right hand bent on uterine body contact.
  Both hands catch utero withdrawal into one on another with arms outstretched. Fixed uterus right hand, left hand, with levers legs combines lateroflexion-rotation parameters of lumbar spine to improve uterine ligaments stretch, repeat technique to tissue relaxation. Then perform massage-cranial caudo zigzag with anteroposterior thrust. (overall hemodynamic maneuver). Finally do anteroposterior pumping about uterine body generating positive and negative pressures.
  Hand therapist will keep in touch at all times on the suprapubic region of the patient.
  Interventions: Other: Reproductive Technique Gimilio
- Placebo Intervention (Placebo Comparator): The researcher puts his right hand on the right shoulder of the patient for 20 times Metronome.
  Interventions: Other: Placebo Intervention

INTERVENTIONS:
Other: Reproductive Technique Gimilio — Patient supine, legs in triple flexion, feet on table, controlling legs left hand and right hand bent on uterine body contact.
  Both hands catch utero withdrawal into one on another with arms outstretched. Fixed uterus right hand, left hand, with levers legs combines lateroflexion-rotation parameters of lumbar spine to improve uterine ligaments stretch, repeat technique to tissue relaxation. Then perform massage-cranial caudo zigzag with anteroposterior thrust. (overall hemodynamic maneuver). Finally do anteroposterior pumping about uterine body generating positive and negative pressures.
  Hand therapist will keep in touch at all times on the suprapubic region of the patient.
  Other Names: Uterine Vascular Technique of Gimilio
  Arms: Reproductive Technique Gimilio
Other: Placebo Intervention — Patient supine, legs in triple flexion, feet on table. Physical Therapist take contact with his right hand in patient's belly for 5 minutes, without any movement.
  Other Names: Placebo Intervention technique
  Arms: Placebo Intervention

SUMMARY:
Ivanovski shows that by studying the vascular impedance can calculate the optimal uterine receptivity in IVF. A reduced vascular resistance and increased blood flow rate improves the chance of pregnancy.

Dr. Luis T. Mercé says: "After evaluating 40 cycles of IVF (In Vitro Fertilization) have found that the pregnancy rates increases with increasing endometrial volume. It has also advocated that the endometrial blood flow better reflects uterine receptivity, since the endometrium is where will take place the embryo implantation. Merce also claims to have found that the pregnancy rate increases with increasing endometrial volume and no pregnancies were achieved with endometrial volume less than 3 ml.

These statements motivate us to perform a research project to monitor changes that occur in the uterine endometrial vascularization and subendomertial vascularization after applying a manual physiotherapic technique in menopausal women.

Various authors report that by osteopathic techniques applied on visceral structures, vascular flow rate of the treated bodies increased.

In the literature there are not articles on the subject at hand, but there are references to the manual techniques in the treatment of women with infertility where they state that the manual action for lymphatic congestion in the pelvic region facilitates pregnancy in women infertile.

The practice of visceral osteopathy offers the possibility of accessing the treatment of uterine functional disorders, as well as structures such as uterine ligaments. They influence the fluidic efficiency of uterine arteriovenous system. According to Salamon E., W. Zhu and Stefano GB., provides enough tools to improve the movement of fluids and uterine vascularization.

DETAILED DESCRIPTION:
Introduction Menopause, mark the end of the reproductive period of women. It is a normal part of aging due to decreased production of estrogen and progesterone, associated with the loss of reproductive capacity, having appeared between 48 and 54 years.

Note the difference between menopause and climateric, being climacteric period when the woman has the disappearance of their reproductive function, as well as changes in the secretion of sex hormones, who determining overall change in the body.

Climateric is a sign within the phenomena occurring during menopause. Menopause is the period from 3 to 5 years with symptoms that reflect the beginning of the cessation of ovarian function and postmenopausal between 7 and 10 years. Found indices FSH (follicle stimulating hormone) elevated in early follicular phase, being> 40 IU / L45, the follicular phase of the cycle is shortened, the levels of estradiol and after inhibin folículoestatina decrease, and luteinizing hormone (LH) also increase, but less so than before. During menopause, the ovarian follicles stop responding to FSH and LH, and estradiol drops below 20 pg / mL. Progesterone is clinically undetectable and no disappear menstruation. Hypoestrogenemia, that is the deficit of estrogen levels below 20 pg / ml occurs. The postmenopausal ovary is not an inactive body as it continues to produce both estrogen and androstenedione, although in minimal amounts. Clinical studies suggest that 20 to 50% of postmenopausal women has estrogen levels indicative of follicular activity during the first 6-12 months after the cessation of menstruation.

HYPOTHESIS AND OBJECTIVES

-Hypothesis: Physiotherapy manual techniques improves the uterine vascularization.

-Objectives:

Fundamental objective:

• Quantify the changes that occur in the vascularization index (IV)

Secondary objectives:

* Quantify the changes that occur in vascular indices of endometrial and subendometrial flow Doppler angiography, after running the physiotherapy technique.
* Quantify the changes occurring in the flow rate of the uterine artery (right and left), both before and after running the physiotherapy technique.
* Quantify the longitudinal vascularization measure endometrial / subendometrial and valuing amount of endometrial / subendometrial, both before and after the physiotherapy technique.
* Measure by 3D ultrasound of total uterine volume, both before and after running the physiotherapy technique.

PATIENTS AND METHODS The study population will be infertile women with hypoestrogenemia.

Inclusion criteria:

* Women with hypoestrogenemia and menopausia, being estrogen levels below 20 pg / ml (demonstrated by hormone analysis).
* Women with morphologically normal uterus.
* Women without hormonal treatment of any kind.

Exclusion criteria:

* Patients with any disease in which manipulative therapy is contraindicated. (Contraindicated in the description of the technique)
* Patients with obesity IMC≥30 kg / m2.
* High pain to abdominal palpation.
* Pregnant patients.
* Patients with bleeding disorders.

Sample size:

Given that the primary endpoint of the study is the histogram vascularization index, and according to the estimate by the statistic department of the IVI, the "n" of the study is 52 patients.

All patients are one-sided test for paired samples t. The level of significance is 95% and 80% power.

ANALYSIS:

The results are presented in Excel tables of continuous data, means and standard deviations, which will be interpreted by Dr. Garrido, a member of the research team in charge of statistical analysis.

Methodology Study Design: Prospective experimental intervention study, double blind, paired samples in order to determine the benefit of a medical application technique.

Work plan:

1. Recruitment of patients
2. Study of basal uterine vascularization by Doppler ultrasound prior of the osteopathic technique. The application of ultrasound technique will always performed by the same specialist gynecologist of Doppler (VSS) ultrasound. The scanner is calibrated so that all women are valued with the same calibration.
3. Conducting osteopathic technique. The technique of stretching of the uterine ligaments externally and the rest of the technique together in one technique and applied in a single clinical session will be held. The duration of the execution of the technique, as proposed, will be 30 minutes.
4. Re-evaluation of the uterine vascularization by ultrasound-Doppler after the osteopathic technique. Ultrasound measured is performed within 5 minutes after the execution of the physiotherapeutical technique.
5. Interpretation, with 4DView profram VOCAL, of the obtained volumes of measuring uterine endometrial vascular.
6. Statistical analysis of the data

COSTS OF STUDY:

The research is sponsored by the Juana Crespo's Clinic, so that all costs of patient recruitment and application of diagnostic techniques do not entail direct expenditure on research.

TECHNICAL DESCRIPTION OF ULTRASOUND:

The Doppler application of ultrasound, is an special ultrasound that measures the direction and speed of blood cells as they move through vessels. The movement of blood cells causes a change in pitch of the reflected sound waves (called the Doppler effect). A computer collects and processes the sounds and creates graphs or color pictures that represent the flow through blood vessels.

There is now a new diagnostic methodology, multiplanar volumetric three-dimensional ultrasound technique. This new method, using the available computing resources, allows the observation in different spatial planes (axial, sagittal and coronal) from obtaining volumes of anatomical structures, being the closest thing to a nuclear magnetic resonance (NMR) and facilitating the exploration in two stages, where first is done catch volumes and, in a second time, would be processed and report, it does not require that the probe is connected to be a (4D-View) program that allows working on the data from the computer. Therefore, these new diagnostic techniques using ultrasound Doppler will serve to objectify the potential benefits of the osteopathic techniques.

The ultrasound technique that will be used for the diagnosis of the uterine vascularization is:

1. study using colored transvaginal Doppler ultrasound of right and left uterine arteries, for measuring the resistance index (RI), pulsatility index (PI), peak systolic flow velocity (PSV), flow rate end-diastolic (EDV) and the maximum flow rate (TAmax: time Averaged Maximum Velocity) (these last three parameters after correction of the angle of incidence between the beam and uterine artery Doppler).
2. Multiplanar Ultrasound 3D and three-dimensional ultrasound angiography (powerDoppler) next to the Quick Tools VOCAL (Virtual OrganComputer-AidedAnalysis), for the study of endometrial volume and rates of endometrial vascularization and subendometrial generated from the histogram data of angiography 3D Doppler.

   * Index Vascularization (IV).
   * Index Flow (IF).
   * index Vascularization flow (IFV).

Three-dimensional ultrasound is equipped with a computer software to measure the volumes generated waves. The best known and reported program is called VOCAL, an acronym derived from the first letters of the English words Virtual Organ Computer-aided Analysis. Not with standing the VOCAL acronyms it can also be interpreted as calculation of volume, VOlumeCALculation Saxon words. This method allows to delimit the volumes of a region of interest using a rotational method.

We will use Doppler ultrasound, transvaginal application to assess the following variables:

* Primary variable (or dependent):

  -Endometrial/subendometrial Vascularization Index (VI).
* Explanatory variables that could change or influence the behavior of key variables are included in the exclusion criteria.
* Control variables (dependent):
* Resistance index (RI) of both uterine arteries. It is an independent measurement of the angle of the ultrasound beam. It is calculated as:
* pulsatility index (IP) of both uterine arteries.
* Average maximum flow rate (TAmax) of both uterine arteries. Angle correction required.
* peak systolic velocity (PSV) and end diastolic velocity (EDV) of both uterine arteries. Angle correction required.
* endometrial / subendometrial vascular map, evaluated qualitatively: the absence / presence of vessels.
* endometrial volume obtained with the VOCAL application from multiplanar sections of the uterus.
* Histogram of 3D angiography:

  * Index Of endometrial and subendometrial flow (IF).
  * Index Vascular flow (IFV).

DESCRIPTION PHYSIOTHERAPEUTICAL MANUAL TECHNIQUE The place where the event will take will be a table equipped with the ultrasound equipement and prepared for measurement, always accompanied by the same sonographer gynecologist, for all women involved in the study.

With the patient supine and lower limb triple flexion resting your feet on the table, put the left hand controlling the bent legs and the right hand, having caught a fold of skin, making contact on the uterine body. Both hands caught withdrawal into the uterine body, one on one with the right arm fixed extendidos. Right hand in uterus, while the left hand, with the levers of the lower limbs, combine parameters lateroflexion-rotation of the lumbar spine for improve stretching the uterine ligaments, repeating the movement until tissue relaxation. Subsequently we conducted a zigzag caudo-cranial massage anteroposterior making a push (Global hemodynamic maneuver) and finally we carried out an anteroposterior pumping on the uterine body generating positive and negative pressures.

The therapist's hand will keep in touch at all times on the suprapubic region of the patient.

ELIGIBILITY:
Inclusion criteria:

* Women with hypoestrogenemia and menopausia, being estrogen levels below 20 pg / ml (demonstrated by hormone analysis).
* Women with morphologically normal uterus.
* Women without hormonal treatment of any kind.

Exclusion criteria:

* Patients with any disease in which manipulative therapy is contraindicated. (Contraindicated in the description of the technique)
* Patients with obesity IMC≥30 kg / m2.
* High pain to abdominal palpation.
* Pregnant patients.
* Patients with bleeding disorders.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Increased uterine vascular flow after application of the Reproductive Physioterapeutic Technique. | 5 minutes after application of Reproductive Therapy Technique Gimilio

CONTACTS AND LOCATIONS:
Overall Officials: César M Gimilio Martínez, D., Principal Investigator — University of Valencia
Locations (1):
- Catholic University of Valencia, Torrent, Valencia, Spain

REFERENCES:
- [Background] Jones HW Jr, Cooke I, Kempers R, Brinsden P, Saunders D. International Federation of Fertility Societies Surveillance 2010: preface. Fertil Steril. 2011 Feb;95(2):491. doi: 10.1016/j.fertnstert.2010.08.011. PMID 20813358
- [Background] Faddy MJ, Gosden RG, Gougeon A, Richardson SJ, Nelson JF. Accelerated disappearance of ovarian follicles in mid-life: implications for forecasting menopause. Hum Reprod. 1992 Nov;7(10):1342-6. doi: 10.1093/oxfordjournals.humrep.a137570. PMID 1291557
- [Background] Budak E, Garrido N, Soares SR, Melo MA, Meseguer M, Pellicer A, Remohi J. Improvements achieved in an oocyte donation program over a 10-year period: sequential increase in implantation and pregnancy rates and decrease in high-order multiple pregnancies. Fertil Steril. 2007 Aug;88(2):342-9. doi: 10.1016/j.fertnstert.2006.11.118. Epub 2007 Feb 28. PMID 17335819
- [Background] Remohi J, Gallardo E, Guanes PP, Simon C, Pellicer A. Donor-recipient synchronization and the use of gonadotrophin-releasing hormone agonists to avoid the premature luteinizing hormone surge in oocyte donation. Hum Reprod. 1995 Dec;10 Suppl 2:84-90. doi: 10.1093/humrep/10.suppl_2.84. PMID 8745305
- [Background] El-Mazny A, Abou-Salem N, Elshenoufy H. Three-dimensional power Doppler study of endometrial and subendometrial microvascularization in women with intrauterine device-induced menorrhagia. Fertil Steril. 2013 Jun;99(7):1912-5. doi: 10.1016/j.fertnstert.2013.01.151. Epub 2013 Mar 7. PMID 23465819
- [Background] Wurn BF, Wurn LJ, King CR, Heuer MA, Roscow AS, Scharf ES, Shuster JJ. Treating female infertility and improving IVF pregnancy rates with a manual physical therapy technique. MedGenMed. 2004 Jun 18;6(2):51. PMID 15266276
- [Background] Mercier J, Miller K. Mercier therapy helps infertile women achieve pregnancy. Midwifery Today Int Midwife. 2013 Spring;(105):40, 68. No abstract available. PMID 23581202
- [Background] Nelson KE, Sergueef N, Glonek T. The effect of an alternative medical procedure upon low-frequency oscillations in cutaneous blood flow velocity. J Manipulative Physiol Ther. 2006 Oct;29(8):626-36. doi: 10.1016/j.jmpt.2006.08.007. PMID 17045096
- [Background] Ivanovski M, Damcevski N, Radevska B, Doicev G. Assessment of uterine artery and arcuate artery blood flow by transvaginal color Doppler ultrasound on the day of human chorionic gonadotropin administration as predictors of pregnancy in an in vitro fertilization program. Akush Ginekol (Sofiia). 2012;51(2):55-60. PMID 23234017
- [Background] Raine-Fenning NJ, Campbell BK, Clewes JS, Kendall NR, Johnson IR. The reliability of virtual organ computer-aided analysis (VOCAL) for the semiquantification of ovarian, endometrial and subendometrial perfusion. Ultrasound Obstet Gynecol. 2003 Dec;22(6):633-9. doi: 10.1002/uog.923. PMID 14689538
- [Background] Ely JW, Kennedy CM, Clark EC, Bowdler NC. Abnormal uterine bleeding: a management algorithm. J Am Board Fam Med. 2006 Nov-Dec;19(6):590-602. doi: 10.3122/jabfm.19.6.590. PMID 17090792
- [Background] Maulik D, Yarlagadda P, Youngblood JP, Ciston P. Comparative efficacy of umbilical arterial Doppler indices for predicting adverse perinatal outcome. Am J Obstet Gynecol. 1991 Jun;164(6 Pt 1):1434-9; discussion 1439-40. doi: 10.1016/0002-9378(91)91421-r. PMID 2048589
- [Background] Erskine RL, Ritchie JW. Umbilical artery blood flow characteristics in normal and growth-retarded fetuses. Br J Obstet Gynaecol. 1985 Jun;92(6):605-10. doi: 10.1111/j.1471-0528.1985.tb01399.x. PMID 4005201
- [Background] Koster K, Poulsen Nautrup C, Gunzel-Apel AR. A Doppler ultrasonographic study of cyclic changes of ovarian perfusion in the Beagle bitch. Reproduction. 2001 Sep;122(3):453-61. doi: 10.1530/rep.0.1220453. PMID 11597310
- [Background] Oldenhave A, Netelenbos C. Pathogenesis of climacteric complaints: ready for the change? Lancet. 1994 Mar 12;343(8898):649-53. doi: 10.1016/s0140-6736(94)92641-7. No abstract available. PMID 7906816
- [Background] Khaw KT. Epidemiology of the menopause. Br Med Bull. 1992 Apr;48(2):249-61. doi: 10.1093/oxfordjournals.bmb.a072546. PMID 1450870
- [Background] Grattarola R, Secreto G, Recchione C. Correlation between urinary testosterone or estrogen excretion levels and interstitial cell-stimulating hormone concentrations in normal postmenopausal women. Am J Obstet Gynecol. 1975 Feb 1;121(3):380-1. doi: 10.1016/0002-9378(75)90016-2. PMID 1115152
- [Background] Gambrell RD Jr. The menopause: benefits and risks of estrogen-progestogen replacement therapy. Fertil Steril. 1982 Apr;37(4):457-74. doi: 10.1016/s0015-0282(16)46149-2. PMID 7040116
- [Background] Ng EH, Chan CC, Tang OS, Yeung WS, Ho PC. Changes in endometrial and subendometrial blood flow in IVF. Reprod Biomed Online. 2009 Feb;18(2):269-75. doi: 10.1016/s1472-6483(10)60265-9. PMID 19192349